CLINICAL TRIAL: NCT06686511
Title: The Effect of Preoperative Counseling on Emergence Agitation in Patients Candidate for Nasal Surgeries : a Prospective Randomized Controlled Study
Brief Title: The Effect of Preoperative Counseling on Emergence Agitation in Patients Candidate for Nasal Surgeries
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Maged Abdel-Wahab Abdel-Aziz, pricipal investigator, Cairo University
Other Study IDs: counseling and agitation
Record Dates: First submitted 2024-10-28; First posted 2024-11-13 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Postoperative Agitation
Keywords: agitation; counseling; nasal surgeries
MeSH Terms: conditions — Psychomotor Agitation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- - Group A: Will ask them to close their nose completely by their hands and take their breath only from the mouth for 2 to 3 minutes before induction of GA.
  : immediately after extubation we will tell them many times at their ear that the operation has been finished and ask them to take their breath from the mouth as they counselled and trained at preoperative period
- ● Group B: Will start the induction of anesthesia without any preoperative counselling of nasal closure .
  this group will undergo extubation and should be instructed to use their nose for breathing without Without preoperative counselling

SUMMARY:
Emergence agitation is a post anesthetic phenomenon that develops in the early phase of general anesthesia recovery,The aim of our study to investigate the effect of preoperative educational counselling of the patient undergoing nasal surgery on emergence agitation .

DETAILED DESCRIPTION:
While its pathogenesis remains unclear, previous studies reported that ENT (ear, nose, and throat) surgical procedures have a higher incidence of emergence agitation in both adults and children. Especially, our clinical impression is that nasal surgical patients admitted to the postbanesthesia care unit (PACU) have suffered emergence agitation more frequently than other surgical patients, possibly due to a sense of suffocation during emergence from anesthesia.

preoperative counselling and repeated verbal stimulation of orientation may serve as a simple and easily applicable strategy to reduce emergence agitation after general anaesthesia .

There have been studies looking into the effect of pre-operative counselling on individual aspects internationally like anxiety, BMI, serum cholesterol , length of stay , pain .( Six trials were identified and have produced conflicting findings. Some trials have demonstrated the effects of preoperative education on improving physical and psychosocial recovery of cardiac patients, while others found no evidence that patients' anxiety is reduced or of any effect on pain or hospital stay) .

To our knowledge there was no study investigating the impact of preoperative counselling on postoperative agitation following nasal surgeries, The aim of our study to investigate the effect of preoperative educational counselling of the patient undergoing nasal surgery on emergence agitation .

ELIGIBILITY:
Inclusion Criteria:

* Both genders.
* Patients undergoing nasal surgery
* American Society of Anesthesiologist (ASA) I or II physical status.
* Between 18 and 65 years of age.

Exclusion Criteria:

* ● Patients with communication difficulties.

  * ASA Ⅲ and Ⅳ patients.
  * Mentally retarded patients.
  * In-ability to postpone anti-coagulation medications.
  * Central or peripheral neurological disease.
  * Drug or alcohol abuse.
  * Localized infection at nose.
  * Bleeding disorder (platelets count less than 100,000 or INR more than 1.4)

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ASA I or II patients of both genders undergoing nasal surgery in the age between 21 to 65 years old will be included in the study
Sampling Method: Probability Sample
Enrollment: 256 (Actual)
Dates: Start 2024-11-25 (Actual); Primary Completion 2025-10-25 (Actual); Study Completion 2025-11-15 (Actual)

PRIMARY OUTCOMES:
The incidence of emergence agitation using AONO s scale(percentage of patients having score of 3 or 4) | scale immediately after extubation and then every 5 minutes for 20 minutes
  ● AONO s four point agitation scale The scale is decribed as 1 = calm; 2 = not calm but could be easily calmed; 3 = not easily calmed, moderately agitated or restless; and 4 = combative, excited, or disoriented.

SECONDARY OUTCOMES:
heart rate in beats per minute | immediately after extubation and then every 5 minutes for 20 minutes
systolic blood pressure in mmhg | immediately after extubation and then every 5 minutes for 20 minutes
mean blood pressure in mmhg | immediately after extubation and then every 5 minutes for 20 minutes
oxygen saturation in % | immediately after extubation and then every 5 minutes for 20 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Maged aw el gendy, lecturer, Principal Investigator — kaser al aini cairo university; Maged aw el gendy, lecturer, Principal Investigator — university
Locations (1):
- operating ENT theater kasr alaini hospital, Cairo, Manil, Egypt

IPD SHARING:
Plan to Share IPD: Yes
sharing the results
Supporting Information: Study Protocol, SAP, CSR

REFERENCES:
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/17179249/